CLINICAL TRIAL: NCT02714127
Title: Collection of First-void Urine Samples for the Development of Standard Operating Procedures for Cervical (Pre)Cancer Biomarker Detection in First-void Urine: the BM-SOP Study
Brief Title: Standard Operating Procedures for Cervical (Pre)Cancer Biomarker Detection in First-void Urine (BM-SOP Study)
Acronym: BM-SOP
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Research Foundation Flanders (Other); University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Pierre Van Damme, Professor Pierre Van Damme, MD, PhD, Universiteit Antwerpen
Other Study IDs: B300201525585
Record Dates: First submitted 2016-03-10; First posted 2016-03-21 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Cervical Cancer
Keywords: Human Papillomavirus; Biomarker; Self-sampling; First-void urine; Cervicovaginal fluid; Colposcopy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — First-void urine samples and Cervicovaginal lavage fluid (VagLav) samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Women (25-64 years old) with abnormal cytology results and/or (high risk) HPV infection refered for colposcopy, and hence possibly diagnosed with an (high risk) HPV infection and/or cervical (pre)cancerous lesions.
  No clinical evaluations/interventions will be performed by our research group. Participants have an already scheduled colposcopy exam. However, this visit is not an extra investigation that the participants should undergo when participating in the study.
  Interventions: Other: First-void urine collection; Other: Cervicovaginal lavage fluid collection
- Controls: Healthy women (25-64 years old), falsely diagnosed with abnormal cytology and/or (high risk) HPV infection, but referred for colposcopy, are included as negative controls. Based on a specificity of 76.14% of the HPV type-specific PCR (polymerase chain reaction) used, an estimated 24 out of these 100 participants will be incorrectly scheduled for colposcopy and serve as the control group.
  No clinical evaluations/interventions will be performed by our research group. Participants have an already scheduled colposcopy exam. However, this visit is not an extra investigation that the participants should undergo when participating in the study.
  Interventions: Other: First-void urine collection; Other: Cervicovaginal lavage fluid collection

INTERVENTIONS:
Other: First-void urine collection — One time collection of ca. 20ml of first-void urine (i.e. the initial stream of the urine void) with the Colli-PeeTM device (Novosanis).
  Other Names: FV urine
Other: Cervicovaginal lavage fluid collection — During colposcopy, the cervicovaginal region is rinsed for 2 minutes with 50 ml acetic acid (5%). This fluid is not discarded like it is done usually, but the remaining lavage fluid (5% acetic acid containing cervicovaginal fluid) will be collected.
  Other Names: VagLav

SUMMARY:
The aim of the study is to develop robust analytical protocols for first-void urine sample preparation and biomarker assays to analyze a panel of biomarkers in first-void urine for improved diagnosis of cervical (pre)cancer lesions.

DETAILED DESCRIPTION:
In total 100 women will be included in this trial, women diagnosed with abnormal cytology results and/or high risk HPV (Human Papillomavirus) infection scheduled for a colposcopy exam. These women are asked to collect a first-void urine sample with the Colli-PeeTM device, prior to their colposcopy exam at the clinic. The collected urine samples will be used for the development and optimisation of robust analytical protocols for first-void urine sample preparation and biomarker assays.

During colposcopy, the cervix will be visually inspected, whether or not combined with a biopsy for histological confirmation. Colposcopy is a procedure to identify abnormalities by using a colposcope that gives an illuminated, magnified view of the cervical region. It often includes rinsing the cervicovaginal region with 50 ml acetic acid (5%). Here, this fluid will be collected and serve as the intermediate step between biomarkers in cervicovaginal secretions and urine.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 25-64 year old
* Women scheduled for a colposcopy exam due to abnormal cytology result according to the Bethesda classification 2001 (NILM, AGC (Atypical Glandular Cells), ASC-US (Atypical Squamous Cells of Undetermined Significance), ASC-H (Atypical Squamous Cells - cannot exclude HSIL), LSIL (Low-grade Squamous Intraepithelial Lesion), HSIL (High-grade Squamous Intraepithelial Lesion), invasive carcinoma), and/or positive for hrHPV infection. NILM (Negative for Intraepithelial Lesion or Malignancy) are only included when positive for hrHPV infection.
* Signing informed consent form (ICF).
* Giving consent to the research team (CEV) to contact his/her general practioner and/or gynaecologist to access details of the participants HPV vaccination (schedule) and results of cervical smears/cytology, HPV tests, colposcopy, and biopsy (included in ICF).

Exclusion Criteria:

* Participating in another clinical study at the same time of participating in this study.
* Not able to understand the information brochure/what the study is about.
* Anything in the opinion of the investigator that would prevent volunteers from completing the study or put the volunteer at risk.

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The cohort of women involves 100 women, diagnosed with an abnormal smear and/or high risk HPV infection (cytology results already available) requested for colposcopic examination. During this colposcopic examination, cervical samples are collected and send to the pathology laboratory. In addition, these women are asked to collect a first-void urine sample with the Colli-PeeTM device and fill in a questionnaire, prior to their colposcopy exam at the clinic (UZA), during which a cervicovaginal lavage fluid sample will be collected as well.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Concentration of cervical cancer biomarkers in first-void urine | Within 6 months after study completion
  To detect candidate biomarkers (originally identified in cervical cells, tissue biopsies, and cervicovaginal fluid (CVF); HPV DNA type(s), viral load (copies/cel), proteins, (m)RNA, methylated (HPV and human) DNA, immunoglobulins; in first-void urine samples from 100 women scheduled for colposcopy due to abnormal cytology.

SECONDARY OUTCOMES:
Preference of women for self-sampling methods | Within 6 months after study completion
  Gather information about the preference of women for first-void urine sample collection compared to the currently available self-sampling methods, and a clinician collected sample (smear).
Concentration of cervical cancer biomarkers in VagLav samples versus first-void urine | Within 6 months after study completion
  To compare the presence of candidate biomarkers (originally identified in cervical cells, tissue biopsies, and cervicovaginal fluid (CVF); HPV DNA type(s), viral load (copies/cel), proteins, (m)RNA, methylated (HPV and human) DNA, immunoglobulins; in paired first-void urine and VagLav samples from 100 women scheduled for colposcopy due to abnormal cytology.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Van Damme, Prof MD PhD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Wiebren Tjalma, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No